CLINICAL TRIAL: NCT02568267
Title: An Open-Label, Multicenter, Global Phase 2 Basket Study of Entrectinib for the Treatment of Patients With Locally Advanced or Metastatic Solid Tumors That Harbor NTRK1/2/3, ROS1, or ALK Gene Rearrangements
Brief Title: Basket Study of Entrectinib (RXDX-101) for the Treatment of Patients With Solid Tumors Harboring NTRK 1/2/3 (Trk A/B/C), ROS1, or ALK Gene Rearrangements (Fusions)
Acronym: STARTRK-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-101-02; 2015-003385-84 (EudraCT Number); GO40782 (Other: Hoffman-La Roche)
Expanded Access: NCT03066661 (No longer available)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Cholangiocarcinoma; Colorectal Cancer; Head and Neck Neoplasms; Lymphoma, Large-Cell, Anaplastic; Melanoma; Neuroendocrine Tumors; Non-Small Cell Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Papillary Thyroid Cancer; Primary Brain Tumors; Renal Cell Carcinoma; Sarcomas; Salivary Gland Cancers; Adult Solid Tumor
Keywords: Entrectinib; RXDX-101; TrkA; TrkB; TrkC; NTRK1; NTRK2; NTRK3; ROS1; ALK; Trk Fusions; NTRK Gene Rearrangements; ROS1 Fusions; ROS1 Gene Rearrangements; ALK Fusions; ALK Gene Rearrangements; Basket study; Non-small cell lung cancer; Colorectal cancer; Salivary gland cancers; Primary brain tumors; Melanoma; Sarcomas; Papillary thyroid cancer; Renal cell cancer; Pancreatic cancer; Breast cancer; Cholangiocarcinoma; Head & Neck cancers; Ovarian cancer; Neuroendocrine tumors
MeSH Terms: conditions — Breast Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Head and Neck Neoplasms; Lymphoma, Large-Cell, Anaplastic; Melanoma; Neuroendocrine Tumors; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Neoplasms; Thyroid Cancer, Papillary; Brain Neoplasms; Carcinoma, Renal Cell; Sarcoma; Salivary Gland Neoplasms | interventions — entrectinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- NTRK1/2/3-rearranged NSCLC (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ROS1-rearranged NSCLC (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ALK- or ROS1-rearranged NSCLC (Experimental): with CNS-only progression previously treated with crizotinib (NOTE: The ALK-rearranged portion of this arm is now closed to enrollment.)
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- NTRK/1/2/3-rearranged mCRC (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ROS1-rearranged mCRC (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ALK-rearranged mCRC (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- NTRK1/2/3-rearranged other solid tumor (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ROS1-rearranged other solid tumor (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- ALK-rearranged other solid tumor (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib

INTERVENTIONS:
Drug: Entrectinib — TrkA/B/C, ROS1, and ALK inhibitor
  Other Names: RXDX-101

SUMMARY:
This is an open-label, multicenter, global Phase 2 basket study of entrectinib (RXDX-101) for the treatment of patients with solid tumors that harbor an NTRK1/2/3, ROS1, or ALK gene fusion. Patients will be assigned to different baskets according to tumor type and gene fusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of locally advanced or metastatic solid tumor that harbors an NTRK1/2/3, ROS1, or ALK gene rearrangement
* For patients enrolled via local molecular testing, an archival or fresh tumor tissue (unless medically contraindicated) is required to be submitted for independent central molecular testing at Ignyta's CLIA laboratory post-enrollment
* Measurable or evaluable disease
* Patients with CNS involvement, including leptomeningeal carcinomatosis, which is either asymptomatic or previously-treated and controlled, are allowed
* Prior anticancer therapy is allowed (excluding approved or investigational Trk, ROS1, or ALK inhibitors in patients who have tumors that harbor those respective gene rearrangements)

  - Note: prior treatment with crizotinib is permitted only in ALK- or ROS1-rearranged NSCLC patients presenting with CNS-only progression. Other ALK inhibitors are prohibited.
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed after prior chemotherapy or small molecule targeted therapy
* At least 4 weeks must have elapsed since completion of antibody-directed therapy
* Prior radiotherapy is allowed if more than 14 days have elapsed since the end of treatment
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and minimum life expectancy of 4 weeks
* Adequate organ function as defined per protocol
* Ability to swallow entrectinib intact
* Other protocol specified criteria

Exclusion Criteria:

* Current participation in another therapeutic clinical trial
* Prior treatment with approved or investigational Trk, ROS1, or ALK inhibitors in patients who have tumors that harbor those respective gene rearrangements

  - Note: prior treatment with crizotinib is permitted only in ALK- or ROS1-rearranged NSCLC patients presenting with CNS-only progression. Other ALK inhibitors are prohibited.
* History of other previous cancer that would interfere with the determination of safety or efficacy
* Familial or personal history of congenital bone disorders, or bone metabolism alterations
* Incomplete recovery from any surgery
* History of recent (within the past 3 months) symptomatic congestive heart failure or ejection fraction ≤50% observed during screening for the study
* History of non-pharmacologically induced prolonged QTc interval
* History of additional risk factors for torsades de pointes
* Peripheral neuropathy Grade ≥ 2
* Known active infections
* Active gastrointestinal disease or other malabsorption syndromes
* Known interstitial lung disease, interstitial fibrosis, or history of tyrosine kinase inhibitor-induced pneumonitis
* Other protocol specified criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RECIST v1.1

SECONDARY OUTCOMES:
Duration of Response | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RECIST v1.1
Time to Response | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RECIST v1.1
Clinical Benefit Rate | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RECIST v1.1
Intracranial Tumor Response | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RANO or RANO-BM, as applicable
CNS Progression-free Survival | Approximately 24 months
  Assessed by blinded independent central review (BICR) using RANO or RANO-BM, as applicable
Progression-free Survival | Approximately 30 months
  Assessed by Kaplan-Meier method
Overall Survival | Approximately 36 months
  Assessed by Kaplan-Meier method
Population PK | Approximately 24 months
  Assessed by Kaplan-Meier method
Adverse Events | Approximately 36 months
  Type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities, graded by the NCI CTCAE
Quality of Life | Approximately 24 months
  Assessed with the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) and the Euro-QoL Group EQ-5D. NSCLC and mCRC patients will complete the lung cancer and colorectal cancer specific modules, QLQ-LC13 and QLQ-CR29, respectively
Bone Growth and Bone Mineral Density | Approximately 30 months
  Assessed with DHA scans
Bone Biomarkers | Approximately 30 months
  Measured by blood

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (130):
- United States (53):
  - Dignity Health St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope Cancer Center, Duarte, California
  - City of Hope Duarte - Comprehensive Cancer Center, Investigational Drug Services, Duarte, California
  - Scripps Clinic, La Jolla, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Southern California Kaiser Permanente, Los Angeles, California
  - University of Southern California Medical Center, Los Angeles, California
  - Univ Of California Irvine College Of Medicine, Orange, California
  - UCSF Mount Zion Medical Ctr, San Francisco, California
  - UCSF Mission Bay, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Southeastern Regional Medical Center, Inc., Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Advocate Medical Group - Park Ridge, Luther Lane - Oncology, Park Ridge, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Weinberg Cancer Institution at Franklin Square, Baltimore, Maryland
  - Massachusetts General Hosp CAR, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - North Shore Hem Onc Associates, East Setauket, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - OSU, James Cancer Hospital, Columbus, Ohio
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health & Science Univ, Portland, Oregon
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Norfolk, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria
- Pharmacy, Edegem, Belgium
- China (9):
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Beijing Cancer Hospital, Beijing
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shanghai chest hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shenzhen People's Hospital, Shenzhen
- France (10):
  - Institut de Cancerologie de l Ouest, Angers
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Nord - AP-HM Marseille#, Marseille
  - Institut de Recherche en Cancérologie de Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut De Cancerologie De L'ouest - Rene Gauducheau - Biology, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitaetsmedizin Goettingen, Göttingen
  - NCT Uniklinikum Heidelberg, Heidelberg
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
  - Queen Elizabeth Hospital, Kowloon
  - The Chinese University of Hong Kong, Shatin
- Italy (7):
  - Seconda Università degli Studi di Napoli, Napoli, Campania
  - Università Campus Bio-Medico di Roma, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia, Umbria
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Japan (11):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital, Chūō
  - NHO Kyushu Cancer Center, Fukuoka
  - Hyogo Cancer Center, Dept of Respiratory Medicine, Hyōgo
  - National Cancer Center Hospital, Kashiwa-shi
  - NHO Shikoku Cancer Center, Matsuyama
  - Miyagi Cancer Center, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka City General Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
- Netherlands (2):
  - NKI The Netherlands Cancer Institute, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Gliwice
  - Szpital Kliniczny Przemienienia Panskiego Uni. Medycznego im. Karola Marcinkowskiego, Późna
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Klinika Nowotworow Ukladu Chlonnego, Warsaw
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center., Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (8):
  - Centro Nacional de Investigaciones Oncológicas(CNIO), Fuenlabrada, Madrid
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Sarah Cannon Research Institute, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Desai AV, Bagchi A, Armstrong AE, van Tilburg CM, Basu EM, Robinson GW, Wang H, Casanova M, Andre N, Campbell-Hewson Q, Wu Y, Cardenas A, Ci B, Ryklansky C, Devlin CE, Meneses-Lorente G, Wulff J, Hutchinson KE, Gajjar A, Fox E. Efficacy and safety of entrectinib in children with extracranial solid or central nervous system (CNS) tumours harbouring NTRK or ROS1 fusions. Eur J Cancer. 2025 May 2;220:115308. doi: 10.1016/j.ejca.2025.115308. Epub 2025 Feb 22. PMID 40086048
- [Derived] Choudhury NJ, Jun Woo H, Chen M, Shah R, Donoghue M, Berger M, Drilon A. Serial Cell-Free DNA Sequencing in ROS1 Fusion-Positive Lung Cancers During Treatment With Entrectinib. JCO Precis Oncol. 2024 Jun;8:e2300721. doi: 10.1200/PO.23.00721. PMID 38848521
- [Derived] Yokota T, Yukino H, Doi M, Ohori H. Real-world experience of tropomyosin receptor kinase inhibition with entrectinib in ETV6-NTRK3 positive metastatic salivary secretory carcinoma: A case series. Head Neck. 2023 May;45(5):E10-E15. doi: 10.1002/hed.27346. Epub 2023 Mar 16. PMID 36924196
- [Derived] Sullivan WG, Hatswell AJ. Letter re: 'Intrapatient comparisons of efficacy in a single-arm trial of entrectinib in tumour-agnostic indications'. ESMO Open. 2021 Dec;6(6):100282. doi: 10.1016/j.esmoop.2021.100282. Epub 2021 Oct 28. No abstract available. PMID 34924145
- [Derived] Doebele RC, Perez L, Trinh H, Martinec M, Martina R, Riehl T, Krebs MG, Meropol NJ, Wong WB, Crane G. Comparative effectiveness analysis between entrectinib clinical trial and crizotinib real-world data in ROS1+ NSCLC. J Comp Eff Res. 2021 Dec;10(17):1271-1282. doi: 10.2217/cer-2021-0131. Epub 2021 Aug 24. PMID 34427452
- [Derived] Dziadziuszko R, Krebs MG, De Braud F, Siena S, Drilon A, Doebele RC, Patel MR, Cho BC, Liu SV, Ahn MJ, Chiu CH, Farago AF, Lin CC, Karapetis CS, Li YC, Day BM, Chen D, Wilson TR, Barlesi F. Updated Integrated Analysis of the Efficacy and Safety of Entrectinib in Locally Advanced or Metastatic ROS1 Fusion-Positive Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Apr 10;39(11):1253-1263. doi: 10.1200/JCO.20.03025. Epub 2021 Mar 1. PMID 33646820
- [Derived] Drilon A, Siena S, Dziadziuszko R, Barlesi F, Krebs MG, Shaw AT, de Braud F, Rolfo C, Ahn MJ, Wolf J, Seto T, Cho BC, Patel MR, Chiu CH, John T, Goto K, Karapetis CS, Arkenau HT, Kim SW, Ohe Y, Li YC, Chae YK, Chung CH, Otterson GA, Murakami H, Lin CC, Tan DSW, Prenen H, Riehl T, Chow-Maneval E, Simmons B, Cui N, Johnson A, Eng S, Wilson TR, Doebele RC; trial investigators. Entrectinib in ROS1 fusion-positive non-small-cell lung cancer: integrated analysis of three phase 1-2 trials. Lancet Oncol. 2020 Feb;21(2):261-270. doi: 10.1016/S1470-2045(19)30690-4. Epub 2019 Dec 11. PMID 31838015
- [Derived] Doebele RC, Drilon A, Paz-Ares L, Siena S, Shaw AT, Farago AF, Blakely CM, Seto T, Cho BC, Tosi D, Besse B, Chawla SP, Bazhenova L, Krauss JC, Chae YK, Barve M, Garrido-Laguna I, Liu SV, Conkling P, John T, Fakih M, Sigal D, Loong HH, Buchschacher GL Jr, Garrido P, Nieva J, Steuer C, Overbeck TR, Bowles DW, Fox E, Riehl T, Chow-Maneval E, Simmons B, Cui N, Johnson A, Eng S, Wilson TR, Demetri GD; trial investigators. Entrectinib in patients with advanced or metastatic NTRK fusion-positive solid tumours: integrated analysis of three phase 1-2 trials. Lancet Oncol. 2020 Feb;21(2):271-282. doi: 10.1016/S1470-2045(19)30691-6. Epub 2019 Dec 11. PMID 31838007
- [Derived] Sigal D, Tartar M, Xavier M, Bao F, Foley P, Luo D, Christiansen J, Hornby Z, Maneval EC, Multani P. Activity of Entrectinib in a Patient With the First Reported NTRK Fusion in Neuroendocrine Cancer. J Natl Compr Canc Netw. 2017 Nov;15(11):1317-1322. doi: 10.6004/jnccn.2017.7029. PMID 29118225